CLINICAL TRIAL: NCT02305719
Title: Regional Anesthesia for Thoracoscopic Surgery
Acronym: RATS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Philip Lang, Assistant professor, Ludwig-Maximilians - University of Munich
Other Study IDs: LudwigMaximilians
Record Dates: First submitted 2014-11-28; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Epidural anesthesia: Patients receiving thoracic epidural anesthesia for thoracoscopic surgery. Standard regimen with 8-20 ml Ropivacaine 0,5% in the epidural catheter. Postopertive Ropivacaine 0,2% 6 ml/h via catheter were administered.
- Serratus-anterior-plane-Block: Patients receiving (ultrasound-guided) Serratus-anterior-plane-Block for thoracoscopic surgery.
  Standard regimen up to 20 ml Ropivacaine 0,5%, were installed. Postopertive Ropivacaine 0,2% 6 ml/h via catheter were administered.
- Local infiltration: Patients receiving local infiltration with up to 20 ml Ropivacaine 0,5% for thoracoscopic surgery (at the site of thoracoscopy)

SUMMARY:
Aim of the study is to evaluate different regional anesthesia regimes for thoracoscopic surgery to evaluate their efficiency in (postoperative) pain control.

Three regional anesthesia forms are evaluated: thoracic epidural anesthesia, (ultrasound-guided) serratus-anterior-plane-block an local infiltration with local anesthetic at the site of performing the thoracoscopy.

DETAILED DESCRIPTION:
A prospective evaluation of different regional anesthesia regimes for thoracoscopic surgery to elucidate their efficiency in (postoperative) pain control.

A day before surgery the patients gave their written informed consent to the study.

Patients choose their favorite regional anesthesia out of the following: thoracic epidural anesthesia, (ultrasound-guided) serratus-anterior-plane-block an local infiltration with local anesthetic at the site of performing the thoracoscopy.

In addition a general anesthesia was applied for the surgical procedure. Anesthesia was maintained using propofol and remifentanil. The patients pain score (visual analog scale), consumption of analgesic medication, satisfaction with pain therapy will be obtained one, six, 24 and 48 hours postoperatively.

These prospective evaluation of different regional anesthetic techniques might provide us data to recommend a procedure for thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thoracoscopic surgery
* ASA 1-3

Exclusion Criteria:

* ASA 4 and 5
* Age under 18 and over 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for thoracoscopic surgery ASA 1-3
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain (visual analog scale) | 48 hours postoperative
  the postoperative Pain, evaluated with a visual analog scale (VAS), was obtained in the first 48 hours postoperatively after thoracoscopic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Lang, M.D., Ph. D., Principal Investigator — Attending
Locations (1):
- University Hospital Munich, Marchioninistr. 15, Munich, Germany